CLINICAL TRIAL: NCT01068262
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Odanacatib (MK0822) in Healthy Male and Postmenopausal Female Subjects
Brief Title: Safety and Tolerability of Odanacatib (0822-059)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-059; 2010_508 (Other: Merck); MK-0822-059
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Panel A - Odanacatib (Experimental): Panel A - Healthy male subjects receiving Odanacatib
  Interventions: Drug: Odanacatib
- Panel A - Placebo (Placebo Comparator): Panel A - Healthy male subjects receiving placebo
  Interventions: Drug: Comparator: Placebo
- Panel B - Odanacatib (Experimental): Panel B - Healthy female subjects receiving Odanacatib
  Interventions: Drug: Odanacatib
- Panel B - Placebo (Placebo Comparator): Panel B - Healthy female subjects receiving placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Odanacatib — Oral doses of Odanacatib 50 mg administered once weekly for 4 consecutive weeks
  Other Names: MK0822
  Arms: Panel A - Odanacatib; Panel B - Odanacatib
Drug: Comparator: Placebo — Oral Placebo tablet administered once weekly for 4 consecutive weeks
  Arms: Panel A - Placebo; Panel B - Placebo

SUMMARY:
This study will test the weighted average inhibition of u-NTx/Cre (aminoterminal crosslinked telopeptide of Type 1 collagen) and AUC (0-168 hours) of Odanacatib

ELIGIBILITY:
Inclusion Criteria:

* male subject between the ages of 50 and 75 years; post menopausal female subjects between the ages of 45 and 75 years
* Subject is in good general health
* Subject has no evidence of metabolic bone disorder other than osteopenia or osteoporosis
* Subject is a non-smoker

Exclusion Criteria:

* Subject works night shift and is unable to avoid nightshift work during the study
* Subject has had major surgery, donated blood or participated in another investigational study with in the past 4 weeks
* Subject has a history of stroke, chronic seizures, or major neurological disease
* Subject has a history of cancer
* Subject consumes excessive amounts of alcohol or caffeine

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-12-08 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Anderson MS, Gendrano IN, Liu C, Jeffers S, Mahon C, Mehta A, Mostoller K, Zajic S, Morris D, Lee J, Stoch SA. Odanacatib, a selective cathepsin K inhibitor, demonstrates comparable pharmacodynamics and pharmacokinetics in older men and postmenopausal women. J Clin Endocrinol Metab. 2014 Feb;99(2):552-60. doi: 10.1210/jc.2013-1688. Epub 2013 Nov 25. PMID 24276460

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Males: Odanacatib (Panel A): Healthy male participants randomized to Odanacatib 50 mg tablet administered once weekly (Qw) for 4 consecutive weeks
- Healthy Males: Placebo (Panel A): Healthy male participants randomized to placebo administered Qw for 4 consecutive weeks.
- Healthy Postmenopausal Females: Odanacatib (Panel B): Healthy postmenopausal female participants randomized to Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Healthy Postmenopausal Females: Placebo (Panel B): Healthy postmenopausal female participants randomized to placebo administered Qw for 4 consecutive weeks
Period: Overall Study
Arm/Group | Healthy Males: Odanacatib (Panel A) | Healthy Males: Placebo (Panel A) | Healthy Postmenopausal Females: Odanacatib (Panel B) | Healthy Postmenopausal Females: Placebo (Panel B)
Started | 23 | 9 | 10 | 2
Completed | 20 | 8 | 9 | 2
Not Completed | 3 | 1 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Males: Odanacatib (Panel A): Healthy male participants randomized to Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Total: Total of all reporting groups
Arm/Group | Healthy Males: Odanacatib (Panel A) | Healthy Males: Placebo (Panel A) | Healthy Postmenopausal Females: Odanacatib (Panel B) | Healthy Postmenopausal Females: Placebo (Panel B) | Total
Number analyzed (Participants) | 23 | 9 | 10 | 2 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline age in each of the four study treatment groups and the total study population
  years | 58.35 (6.11) | 56.44 (6.60) | 57.50 (7.59) | 65.00 (14.14) | 58.07 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 10 | 2 | 12
  Male | 23 | 9 | 0 | 0 | 32

OUTCOME MEASURES:

1. Primary Outcome: Weighted Average Inhibition (WAI) of Urine Aminoterminal Crosslinked Telopeptide of Type I Collagen (u-NTx/Cr) After Administration of Odanacatib 50 mg or Placebo Qw for 4 Weeks in Healthy Males and Postmenopausal Females
Description: uNTx/Cr is a biomarker of bone resorption. Urine samples were obtained predose on Day 1 (Baseline) and at various timepoints up to 336 hr postdose on Day 22 (Week 4). Fold change from baseline in time weighted average (TWA) of uNTx/Cr on log scale was analyzed via a linear mixed effect model. All analyses were carried out on the log-fold scale and final results were reported on the original percent scale in WAI after back transformation. The conversion used was weighted average inhibition (WAI) = (1-exp [mean])*100, where the mean was the least squares (LS) mean of log-transformed ratio (TWA/baseline) from the above model.
Time Frame: Baseline to Week 4
Population: The population of male and postmenopausal female participants on Qw treatment with Odanacatib 50 mg for 4 weeks and were compliant with the protocol. The population of male participants on placebo are also included. Postmenopausal females on placebo were not analyzed for WAI due to there being too few participants in this group (N=2).
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent inhibition
Groups:
- Odanacatib (MK-0822) in Males (Panel A): Healthy males received oral doses of Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Placebo in Males (Panel A): Healthy males received oral doses of placebo administered Qw for 4 consecutive weeks
- Odnacatib (MK-0822) in Postmenopausal Females (Panel B): Healthy postmenopausal females received oral doses of Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Placebo in Postmenopausal Females (Panel B): Healthy postmenopausal females received oral doses of placebo administered Qw for 4 consecutive weeks
Arm/Group | Odanacatib (MK-0822) in Males (Panel A) | Placebo in Males (Panel A) | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Placebo in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 8 | 9 | 0
Percent inhibition | 42.8 [35.5 to 49.3] | -26.4 [-48.9 to -7.3] | 42.7 [30.3 to 52.9] |
Statistical Analysis 1: Comparison: Odanacatib (MK-0822) in Males (Panel A) vs Placebo in Males (Panel A); Test type: Superiority or Other; Linear mixed effect model; Back-transformed least squares estimates and confidence intervals from a linear mixed effect model were performed on natural log-transformed values; Mean Difference (Final Values) = 69.2, 90% CI 2-sided [50.9 to 80.2]
Statistical Analysis 2: Comparison: Odanacatib (MK-0822) in Males (Panel A) vs Odnacatib (MK-0822) in Postmenopausal Females (Panel B); Test type: Superiority or Other; Linear mixed effects model; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.1, 90% CI 2-sided [-14.7 to 14.9]

2. Secondary Outcome: Area Under the Curve of Plasma Concentration-time From 0 to 168 Hours (AUC0-168hr) of Odanacatib at Week 4
Description: Blood samples were obtained predose on Day 1 (Baseline) and at various timepoints up to 336 hr postdose on Day 22 (Week 4) to determine the similarity of steady-state AUC0-168 hr of odanacatib 50 mg administered Qw for 4 weeks in healthy males and postmenopausal females. Characterization of AUC0-168hr after administration of the final, Qw dose of Odanacatib 50 mg at steady state is reflective of the clinical dosing interval.
Time Frame: Baseline, Week 4 (1, 2, 6, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours post-dose)
Population: The population of male and postmenopausal female participants who received Qw treatment with Odanacatib 50 mg for 4 weeks and were compliant with the protocol.
Measure: Geometric Mean (95% Confidence Interval); unit: µM·hr
Groups:
- Odanacatib (MK-0822) in Postmenopausal Females (Panel B): Healthy postmenopausal females received oral doses of Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
Arm/Group | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Odanacatib (MK-0822) in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 9
µM·hr | 33.9 [30.1 to 38.2] | 37.9 [31.9 to 45.0]
Statistical Analysis 1: Comparison: Odnacatib (MK-0822) in Postmenopausal Females (Panel B) vs Odanacatib (MK-0822) in Postmenopausal Females (Panel B); Test type: Superiority or Other; Geometric Mean Ratio (GMR); male/female — Hypothesis: Following 4 weeks of Qw oral dosing of Odanacatib 50 mg, there is no clinically important difference in the true GMR (male/postmenopausal female) of the AUC0-168hr. The GMR is contained within the interval (0.4, 2.0); Estimate = 0.90, 90% CI 2-sided [0.75 to 1.07]

3. Secondary Outcome: Overall Maximum Concentration (Cmax) of Odanacatib in Healthy Male and Postmenopausal Female Participants at Week 4
Description: Blood samples were obtained predose on Day 1 (Baseline) and at various timepoints up to 336 hr postdose on Day 22 (Week 4) to determine the similarity of steady-state Cmax of odanacatib 50 mg administered Qw for 4 weeks in healthy males and postmenopausal females.
Time Frame: Baseline, Week 4 (1, 2, 6, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours post-dose)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Odanacatib (MK-0822) in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 9
nM | 379 [350 to 411] | 409 [363 to 461]
Statistical Analysis 1: Comparison: Odnacatib (MK-0822) in Postmenopausal Females (Panel B) vs Odanacatib (MK-0822) in Postmenopausal Females (Panel B); Test type: Superiority or Other; GMR; GMR = 0.93, 90% CI 2-sided [0.82 to 1.04]

4. Secondary Outcome: Concentration of Odanacatib at 168 Hours (C168hr) in Healthy Male and Postmenopausal Female Participants at Week 4
Description: Blood samples were obtained at 168 hours postdose on Day 22 (Week 4) to determine the similarity of steady-state C168hr (trough concentrations) of odanacatib 50 mg administered Qw for 4 weeks in healthy males and postmenopausal females.
Time Frame: Week 4 (168 hours postdose)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Odanacatib (MK-0822) in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 9
nM | 80 [63 to 102] | 85 [59 to 121]
Statistical Analysis 1: Comparison: Odnacatib (MK-0822) in Postmenopausal Females (Panel B) vs Odanacatib (MK-0822) in Postmenopausal Females (Panel B); Test type: Superiority or Other; GMR; Estimate = 0.95, 90% CI 2-sided [0.66 to 1.35]

5. Secondary Outcome: Overall Time to Maximum Concentration (Tmax) of Odanacatib in Healthy Male and Postmenopausal Female Participants at Week 4
Description: Blood samples were obtained predose on Day 1 (Baseline) and at various timepoints up to 336 hr postdose on Day 22 (Week 4) to determine the similarity of steady-state Tmax of odanacatib 50 mg administered Qw for 4 weeks in healthy males and postmenopausal females.
Time Frame: Baseline, Week 4 (1, 2, 6, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Odanacatib (MK-0822) in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 9
hr | 4.0 [2.0 to 24.0] | 6.0 [2.0 to 12.0]

6. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Odanacatib in Healthy Male and Postmenopausal Female Participants at Week 4
Description: Blood samples were obtained predose on Day 1 (Baseline) and at various timepoints up to 336 hr postdose on Day 22 (Week 4) to determine the similarity of the apparent t1/2 of odanacatib 50 mg administered Qw for 4 weeks in healthy males and postmenopausal females. Harmonic mean, jack-knife standard deviation reported for apparent terminal t1/2.
Time Frame: Baseline, Week 4 (1, 2, 6, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours post-dose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Odanacatib (MK-0822) in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 20 | 8
hr | 89.3 (14.6) | 94.7 (20.4)

7. Secondary Outcome: Number of Participants With At Least One Adverse Event (AE) in the Baseline, Treatment, or Post-Treatment Periods
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the SPONSOR's product, is also an AE. The study determined if the number of AEs experienced by participants receiving Odanacatib 50 mg Qw for 4 consecutive weeks was sufficiently low to permit continued clinical investigation. In addition to AEs during the treatment period and post-treatment follow-up period, AEs may have occurred prior to treatment in screened participants as a result of urine and blood sampling at Baseline.
Time Frame: Up to Day 58
Population: All randomized participants who received ≥1 dose of study treatment
Measure: Number; unit: Participants
Groups:
- Postmenopausal Females: Placebo (Panel B): Healthy postmenopausal females received oral doses of placebo administered Qw for 4 consecutive weeks
Arm/Group | Odanacatib (MK-0822) in Males (Panel A) | Placebo in Males (Panel A) | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Postmenopausal Females: Placebo (Panel B)
Number analyzed (Participants) | 23 | 9 | 10 | 2
Participants | 8 | 5 | 7 | 2

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of the SPONSOR's product, is also an AE. The study determined if the number of participants who discontinued treatment with Odanacatib 50 mg Qw for 4 consecutive weeks due to AEs was sufficiently low to permit continued clinical investigation.
Time Frame: Up to Week 4
Population: All randomized participants who received ≥1 dose of study treatment
Measure: Number; unit: Participants
Arm/Group | Odanacatib (MK-0822) in Males (Panel A) | Placebo in Males (Panel A) | Odnacatib (MK-0822) in Postmenopausal Females (Panel B) | Placebo in Postmenopausal Females (Panel B)
Number analyzed (Participants) | 23 | 9 | 10 | 2
Participants | 2 | 0 | 1 | 0

ADVERSE EVENTS:
Groups:
- Healthy Males: Odanacatib 50 mg (Panel A): Healthy male participants randomized to Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Postmenopausal Females: Odanacatib 50 mg (Panel B): Healthy postmenopausal female participants randomized to Odanacatib 50 mg tablet administered Qw for 4 consecutive weeks
- Postmenopausal Females: Placebo (Panel B): Healthy postmenopausal female participants randomized to placebo administered Qw for 4 consecutive weeks
Arm/Group | Healthy Males: Odanacatib 50 mg (Panel A) | Healthy Males: Placebo (Panel A) | Postmenopausal Females: Odanacatib 50 mg (Panel B) | Postmenopausal Females: Placebo (Panel B)
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/9 | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 8/23 | 5/9 | 7/10 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Males: Odanacatib 50 mg (Panel A) (N=23) | Healthy Males: Placebo (Panel A) (N=9) | Postmenopausal Females: Odanacatib 50 mg (Panel B) (N=10) | Postmenopausal Females: Placebo (Panel B) (N=2)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (5) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycotic allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR has the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.